CLINICAL TRIAL: NCT04510428
Title: A Phase II Randomized Placebo-Controlled, Double Blind, Single-Center, Tolerability and Efficacy Clinical Trial of Ocular Surface Immunoglobulin (OSIG) Eye Drops In Patients With Dry Eye Disease
Brief Title: OSIG-eye Drops Treatment for Dry Eye Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study not initiated.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Sandeep Jain, MD, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-0925
Record Dates: First submitted 2020-08-06; First posted 2020-08-12 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OSIG-Eye Drop (Experimental): Ocular Surface Immune Globulin (OSIG) eye drops 4 mg/ml (0.4%) four times a day for 8 weeks
  Interventions: Drug: Ocular Surface Immune Globulin (OSIG)
- Placebo-Eye Drop (Placebo Comparator): Normal Saline Eye Drops (0.9% NaCl) four times a day for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ocular Surface Immune Globulin (OSIG) — Ocular Surface Immune Globulin (OSIG) eye drops 4 mg/ml (0.4%) four times a day for 8 weeks
  Arms: OSIG-Eye Drop
Drug: Placebo — Normal Saline Eye Drops (0.9% NaCl) four times a day for 8 weeks
  Arms: Placebo-Eye Drop

SUMMARY:
The main objective of this study is to assess the clinical and mechanistic effect of using Ocular surface immunoglobulin (OSIG) eye drops for treating Dry Eye Disease. Therefore, the investigator will perform a prospective, phase II, randomized, placebo-controlled, double-masked, tolerability and efficacy clinical trial using OSIG-eye drops in patients with Dry Eye Disease. This clinical trial will be powered to detect efficacy of the treatment.

This will be a Randomized controlled trial, in which a total of 40 subjects will be enrolled at one clinical site. Subjects will be randomly assigned to one of two groups (#1, #2), with 20 subjects per group. One group will be given placebo (Normal saline eye drops) and the other group will be given eye drops containing the study drug (OSIG). Treatment will be for eight weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Able to Sign and date the informed consent form approved by the Institutional Review Board (IRB)
2. ≥ 18 years of age
3. Patient reported dry eye-related ocular symptoms for at least 3 months before the Screening Visit and use or desire to use artificial tears, ointments or dry eye treatments in the 2 weeks preceding the screening visit
4. Women must be post-menopausal ≥ 1 year, or surgically sterilized. If not, a negative urine pregnancy test is required within 14 days of receiving her first dose of test medication (placebo/ study drug) along with definite evidence of contraceptive use during the duration of the study. Women of reproductive age should use a method of birth control that is acceptable to the subject and the study doctor. This may include oral contraceptive pills, birth control implants, barrier methods or abstinence. If a subject mentions she suspects she may be pregnant after being enrolled, another pregnancy test will be administered. If the test is positive, she will be discontinued from the study immediately.
5. Be willing/able to return for all study visits and to follow instructions from the study investigator and his staff

Exclusion Criteria:

1. Inability to provide informed consent.
2. Vulnerable populations, such as neonates, children, prisoners, institutionalized individuals, or others who may be considered vulnerable populations.
3. Contact lens wear within two weeks of baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2024-01-20 (Estimated)

PRIMARY OUTCOMES:
Mean reduction in Epitheliopathy at week 8, compared to day 1 (pre-dose), as measured by corneal staining score using National Eye Institute (NEI) grading scale. | 8 Weeks
  Corneal staining score as measured by Lissamine Green dye staining using National Eye Institute (NEI) grading scale. Dye is applied to each eye and a slit lamp is used to observe corneal staining. NEI scale relies on a chart that divides the cornea into 5 sections and assigns a value from 0 (absent) to 3 (severe) to each section, based on the density of punctate staining, final staining score being the sum of individual section scores with a range of 0 (minimum) -15 (maximum) points. Complete corneal staining clearance with Lissamine dye defined as a score of 0 indicating the best outcome.
Mean reduction in Dry Eye Disease (DED) symptoms as measured by the Ocular surface disease index (OSDI) score at 8 week, compared to day 1 (pre-dose) | 8 Weeks
  Ocular Surface Disease Index (OSDI), a 12-item questionnaire, assesses symptom of ocular irritation in dry eye disease (DED) and how it affects functioning related to vision in the past week. It has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on 0 to 4 scale with 0 being "none of the time" and 4 being "all of the time." OSDI score range from 0-100 with score 0-12 being normal, 13-22 being mild DED, 23-32 being moderate DED, and >33 being severe DED. OSDI=[(sum of scores for questions answered)×100]/[(total questions answered)×4]

OTHER OUTCOMES:
Visual Analog Scale at 8 Weeks (56 Days) | 8 Weeks
  Subjects will assess their tolerance to the administration of the test medication (placebo/ study drug), utilizing a Visual Analog Scale (VAS). The VAS is a 100 mm horizontal line with verbal descriptors at either end. Subjects will place a single slash mark across the horizontal line between the end labeled "completely intolerable" (0 mm) and "easily tolerable" (100mm). The VAS ratings will be completed after administration of the test medication on Day 1 (post-dose), week 4 and week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Jain, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Illinois Eye and Ear Infirmary, University of Illinois, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No